CLINICAL TRIAL: NCT02232893
Title: A Randomized, Double-Blinded, Placebo-Controlled Trial of TU-100 in Patients Undergoing Laparoscopic Colectomy
Brief Title: Effect of TU-100 in Patients Undergoing Laparoscopic Colectomy
Acronym: TU100P2T3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tsumura USA (Industry)
Collaborators: Cato Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TU100P2T3
Record Dates: First submitted 2014-09-03; First posted 2014-09-05 (Estimated); Results first posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Postoperative Ileus
Keywords: Gastrointestinal Quality of Life Index (GIQLI); Postoperative Quality of Life; Abdominal Bloating; Laparoscopic colectomy; Postoperative ileus (POI)
MeSH Terms: interventions — dai-kenchu-to; 12,13-dihydro-N-methyl-6,11,13-trioxo-5H-benzo(4,5)cyclohepta(1,2-b)naphthalen-5,12-imine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Daikenchuto (TU-100) (Experimental): Daikenchuto (TU-100) 5g TID (15g/day)
  Interventions: Drug: Daikenchuto (TU-100)
- Placebo (Placebo Comparator): Placebo TID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Daikenchuto (TU-100) — Subjects will receive 5g TID (15g/day) of TU-100. Dosage form is granule. Subject will take a daily dose divided 3 times per day for 3 days before surgery and for 28 days after surgery.
  Arms: Daikenchuto (TU-100)
Drug: Placebo — Subjects will receive daily dose of TU-100 placebo. Dosage form is granule. Subject will take a daily dose divided 3 times per day for 3 days before surgery and for 28 days after surgery.
  Arms: Placebo

SUMMARY:
TU-100 is a gastrointestinal drug produced from the three botanical raw materials, Asian ginseng, Zanthoxylum fruit (Japanese pepper), and ginger, based on proprietary aqueous decoction and granulation technology. The aim of this study is to assess the effect of TU-100 on post-operative quality of life during the 4 week postoperative period after straight, hand-assisted, or robot-assisted laparoscopic colectomy. Optimal efficacy parameters for subsequent outcome studies also will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age
* Has a current diagnosis of colon cancer, diverticulitis, or benign colonic neoplasm
* Requires straight, hand-assisted, or robot-assisted laparoscopic colectomy
* Requires hospitalization for surgery and recovery

Exclusion Criteria:

* Has been diagnosed with rectal cancer, advanced or metastatic colon cancer, Crohn disease, ulcerative colitis, or volvulus
* Requires resection of rectal lesion
* Has received or is scheduled to receive chemotherapy during the duration of the study
* Is a pregnant or lactating female
* Has diabetic neuropathy
* Has a history or presence of diabetic gastroparesis
* Has a compromised immune system, either from treatment with corticosteroids or other immunosuppressive agent within 2 weeks of surgery or from immunosuppressive disease (e.g., human immunodeficiency virus)
* Has any other serious condition that might adversely affect suitability for participation in this study, such as liver disorder (including alanine aminotransferase or aspartate aminotransferase level greater than 2.5 times the upper limit of normal), kidney disorders, heart failure, blood disorders, or metabolic disorders
* Has a history or presence of interstitial pneumonia
* Has a history of allergic reaction to ginseng, ginger or Zanthoxylum fruit (Japanese pepper)
* Plans to receive any abdominal irradiation
* Is clinically lactose intolerant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2014-09; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Jensen, M.D., M.P.H., Principal Investigator — Colon & Rectal Surgery Associates
Locations (13):
- United States (13):
  - Los Angeles Site, Los Angeles, California
  - Aurora Site, Aurora, Colorado
  - Weston Site, Weston, Florida
  - Atlanta Site, Atlanta, Georgia
  - Chicago Site, Chicago, Illinois
  - Metairie Site, Metairie, Louisiana
  - Burlington, MA Site, Burlington, Massachusetts
  - Coon Rapids Site, Coon Rapids, Minnesota
  - Minneapolis Site, Minneapolis, Minnesota
  - Jackson Site, Jackson, Mississippi
  - Cleveland Site, Cleveland, Ohio
  - Burlington, VT Site, Burlington, Vermont
  - Spokane Site, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was carried out at 16 sites in the United States (US).
Period: Overall Study
Arm/Group | Daikenchuto (TU-100) | Placebo
Started | 35 | 34
Safety Population | 34 (Pts who rec'd at least 1 dose of study drug. All safety analyses performed using this population.) | 32 (Pts who rec'd at least 1 dose of study drug. All safety analyses performed using this population.)
Primary Endpoint Population | 24 (Patients who provided GIQLI scores both at baseline and Visit 4 were analyzed for primary endpoint) | 19 (Patients who provided GIQLI scores both at baseline and Visit 4 were analyzed for primary endpoint)
Completed | 31 | 27
Not Completed | 4 | 7
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Sponsor request early termination | 0 | 1
Not completed — Developed exclusion criteria | 0 | 1
Not completed — Other | 0 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population - patients who were randomized, underwent surgery after randomization, and received at least one dose of study medication. This population was used for all efficacy analyses.
Groups:
- TU-100: TU-100: 5g TID (15g/day)
  TU-100: Subjects will receive 5g TID (15g/day) of TU-100. Dosage form is granule. Subject will take a daily dose for 3 days before surgery and for 28 days after surgery.
- Placebo: Placebo TID
  Placebo: Subjects will receive daily dose of TU-100 placebo. Dosage form is granule. Subject will take a daily dose for 3 days before surgery and for 28 days after surgery.
- Total: Total of all reporting groups
Arm/Group | TU-100 | Placebo | Total
Number analyzed (Participants) | 34 | 31 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (9.76) | 58.4 (12.4) | 58.6 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 16 | 14 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 32 | 30 | 62
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 34 | 31 | 65

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life After Surgery Based on Gastrointestinal Quality of Life Index (GIQLI) Global Score From Baseline to Visit 4.
Description: The primary endpoint was change in The Gastrointestinal Quality of Life Index (GIQLI) global score from baseline to Visit 4 (Day 15 minus baseline). The global score could range from 0 (lowest quality of life) to 144 (highest quality of life). The effect of TU-100 on the change in GIQLI global score from baseline was assessed by using an analysis of covariance (ANCOVA) model with treatment group as a fixed effect and with baseline GIQLI global score, scheduled surgical location in the colon, and solid food before/after the first flatus as covariates.
Time Frame: Baseline and 15 days
Population: Among the ITT population, patients who provided GIQLI scores both at baseline and Visit 4 were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- TU-100: TU-100: 5g TID (15g/day)
  TU-100: Subjects will receive 5g TID (15g/day) of TU-100. Dosage form is granule. Subject will take a daily dose divided 3 times per day for 3 days before surgery and 28 days after surgery.
- Placebo: Placebo TID
  Placebo: Subjects will receive daily dose of TU-100 placebo. Dosage form is granule. Subject will take a daily dose divided 3 times per day for 3 days before surgery and 28 days after surgery.
Arm/Group | TU-100 | Placebo
Number analyzed (Participants) | 24 | 19
score on a scale | -17.20 (2.76) | -10.10 (2.99)
Statistical Analysis 1: Comparison: TU-100 vs Placebo; Test type: Superiority; p > 0.05, ANCOVA

ADVERSE EVENTS:
Time Frame: 2 months
Groups:
- Daikenchuto (TU-100): Daikenchuto (TU-100) 5g TID (15g/day)
  Daikenchuto (TU-100): Subjects will receive 5g TID (15g/day) of TU-100. Dosage form is granule. Subject will take a daily dose divided 3 times per day for 3 days before surgery and 28 days after surgery.
Arm/Group | Daikenchuto (TU-100) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/32
Serious Adverse Events (participants affected / at risk) | 3/34 | 4/32
Other Adverse Events (participants affected / at risk) | 29/34 | 23/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daikenchuto (TU-100) (N=34) | Placebo (N=32)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Post-operative Ileus (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Post-operative Wound Infection (Infections and infestations) | 1 (1) | 0 (0)
Small bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 0 (0) | 1 (1)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daikenchuto (TU-100) (N=34) | Placebo (N=32)
Nausea (Gastrointestinal disorders) | 13 (13) | 13 (13)
Vomiting (Gastrointestinal disorders) | 5 (5) | 5 (5)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 7 (7) | 5 (5)
Incision site pain (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Procedural nausea (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 7 (7) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 3 (3)
Hypotension (Vascular disorders) | 3 (3) | 3 (3)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Bladder Spasm (Renal and urinary disorders) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/93/NCT02232893/Prot_SAP_000.pdf